CLINICAL TRIAL: NCT06664320
Title: Impact of Mild Acute Normovolemic Hemodilution on Pre-bypass Coagulation Function During Cardiac Surgery
Brief Title: Mild ANH on Pre-bypass Coagulation Function During Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KUH1160030-2
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Mitral Regurgitation; Mitral Stenosis; Tricuspid Regurgitation
Keywords: rotational thromboelastometry; cardiac surgery; acute normovolemic hemodilution; hemodilution; coagulation
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis; Tricuspid Valve Insufficiency; Thrombosis | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): patients undergoing cardiac surgery supposed not to get aucte normovolemic hemodilution (ANH) before CPB
- Acute normovolemic hemodilution group (Active Comparator): patients undergoing cardiac surgery supposed to get aucte normovolemic hemodilution (ANH) before CPB
  Interventions: Procedure: Acute normovolemic hemodilution (ANH); Drug: hydroxyethyl starch (HES 130/0.6)

INTERVENTIONS:
Procedure: Acute normovolemic hemodilution (ANH) — applying acute normovolemic hemodilution (ANH) by using HES 130/0.4 of 5 ml/kg before the initiation of cardiopulmonary bypass
  Arms: Acute normovolemic hemodilution group
Drug: hydroxyethyl starch (HES 130/0.6) — hydroxyethyl starch (HES 130/0.6)
  Arms: Acute normovolemic hemodilution group

SUMMARY:
The impact of acute normovolemic hemodilution (ANH) using hydroxyethyl starch before initiating cardiopulmonary bypass (CPB) on whole blood viscoelastic profile after CPB has not been well established. Patients undergoing cardiac surgery employing moderate hypothermic CPB are randomly allocated into one of two groups: in Group-ANH, ANH is applied by using a balanced hydroxyethyl starch (HES 130/0.6); and in Group-C, ANH is not applied. After weaning from CPB, intergroup differences of INTEM, EXTEM, FIBTEM, and APTEM profiles are analyzed. As a primary outcome, the inter-group differences between maximal clot firmness of EXTEM will be determined at 10 min after ANH in Group-ANH and that at control.

DETAILED DESCRIPTION:
Background: The impact of acute normovolemic hemodilution (ANH) using hydroxyethyl starch before initiating cardiopulmonary bypass (CPB) on whole blood viscoelastic profile after CPB has not been well established. Method: Patients undergoing cardiac surgery employing moderate hypothermic CPB are randomly allocated into one of two groups: in Group-ANH(n=29), ANH is applied by using a balanced hydroxyethyl starch (HES 130/0.6); and in Group-C ANH (n=29)is not applied. Intergroup differences of INTEM, EXTEM, FIBTEM, and APTEM profiles are analyzed. after anesthesia induction (control) and after weaning from CPB and protamine neutralization (after-CPB) in both groups. In Group-ANH, those are determined after ANH (after-ANH). As a primary outcome, the inter-group difference between maximal clot firmness of EXTEM is determined at 10 min after ANH in Group-ANH and that at control. As secondary outcomes, intergroup differences of Hematocrit (Hct), Na+, K+, HCO3-, Ca2+, osmolarity, and s-Cr are determined Intergroup differences of data at T2 are performed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery with cardiopulmonary bypass who signed written informed consent

Exclusion Criteria:

* preoperative renal failure requiring reran replacement therapy
* preoperative liver disease
* preoperative low cardiac output (EF < 50%)
* Preoperative IABP application, Atrial fibrillation, Pacemaker
* contraindication for applying TEE
* intraoperative withdrawal

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximal clot firmness of EXTEM | 10 min after completion of acute normovolemic hemodilution (ANH)
  Maxiaml clot firmess (MCF) of EXTEM of rotational thromboleastometry

SECONDARY OUTCOMES:
Clot formation time of EXTEM | 10 min after completion of acute normovolemic hemodilution
  Clot formation time of EXTEM of rotational thromboleastometry
A10 of FIBTEM | 10 min after completion of acute normovolemic hemodilution
  A10 of FIBTEM of rotational thromboelastometry

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk University Medical Center
Locations (2):
- South Korea (2):
  - Konkuk University Medical Center, Seoul, Seoul
  - Konkuk University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided